CLINICAL TRIAL: NCT02272361
Title: Randomized Controlled Trial Comparing Laparoscopic Sacropexy and Vaginal Mesh Surgery for Women Cystocele Repair: Functional and Anatomical Results at Four Years Follow-up
Brief Title: Trial Comparing Laparoscopic Sacropexy and Vaginal Mesh Surgery for Women Cystocele Repair.
Acronym: PROSPERE4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014_03; 2014-A00258-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Cystocele
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic sacrocolpopexy (Other): laparoscopic sacrocolpopexy
  Interventions: Other: laparoscopic sacrocolpopexy
- vaginal mesh surgery (Other): vaginal mesh surgery
  Interventions: Other: vaginal mesh surgery

INTERVENTIONS:
Other: laparoscopic sacrocolpopexy
  Arms: laparoscopic sacrocolpopexy
Other: vaginal mesh surgery
  Arms: vaginal mesh surgery

SUMMARY:
The primary objective of this study is to compare with PFDI-20 questionnaire the functional outcome of laparoscopic sacrocolpopexy and vaginal mesh surgery in the treatment of symptomatic exteriorised cystocele up to 4 years after surgery.

The secondary objectives of this study are the following:

1. to compare the two techniques for anatomical results based on the clinical evaluation of patients with POP-Q.
2. to overall quality of life assessment and expectations of patients.
3. to compare the two techniques for the long-term safety. The evaluation will focus on the adverse effects of long-term sexual and genital symptoms, urinary and digestive functional symptoms, and chronic pelvic pain.
4. to compare the improvement of the functional outcome assessed by PFDI-20 questionnaire (matched-analysis before versus after).

ELIGIBILITY:
Inclusion Criteria:

* All the patients included in the PROSPERE study will be included in the PROSPERE-4 study. The inclusion criterias for the PROSPERE study are:
* Written informed consent
* insured under the French social security system

Exclusion Criteria:

* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol
* Participation in another trial

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
PFDI-20 score | 4 years
  The patient-reported outcome of the intervention will be evaluated using the symptom score calculated using the PFDI-20. It is a self-administered questionnaire on symptoms of prolapse

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe LUCOT, MD,, Principal Investigator — University Hospital, Lille
Locations (12):
- France (12):
  - Sébatien BLANC, Annecy
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - GCS Flandre Maritime, Grande-Synthe
  - CH La Rochelle Service de Gynécologie Obstétrique, La Rochelle
  - Hôpital BICETRE / Service de Gynécologie Obstétrique, Le Kremlin-Bicêtre
  - CHRU de Lille - Service de Gynécologie médico chirurgicale, Lille
  - CHU de Nîmes, Nîmes
  - Groupe Hospitalier Diaconesses Croix St-Simon, Paris
  - CHI Poissy-St-Germain / Service de gynécologie, Poissy
  - CHU de Poitiers, Poitiers
  - Hôpital de Hautepierre, Strasbourg

REFERENCES:
- [Background] Lucot JP, Fritel X, Debodinance P, Bader G, Cosson M, Giraudet G, Collinet P, Rubod C, Fernandez H, Fournet S, Lesavre M, Deffieux X, Faivre E, Trichot C, Demoulin G, Jacquetin B, Savary D, Botchorichvili R, Campagne Loiseau S, Salet-Lizee D, Villet R, Gadonneix P, Delporte P, Ferry P, Aucouturier JS, Thirouard Y, de Tayrac R, Fatton B, Wagner L, Nadeau C, Wattiez A, Garbin O, Youssef Azer Akladios C, Thoma V, Baulon Thaveau E, Saussine C, Hermieu JF, Delmas V, Blanc S, Tardif D, Fauconnier A; GROG (groupe de recherche en gynecologie et obstetrique). [PROSPERE randomized controlled trial: laparoscopic sacropexy versus vaginal mesh for cystocele POP repair]. J Gynecol Obstet Biol Reprod (Paris). 2013 Jun;42(4):334-41. doi: 10.1016/j.jgyn.2013.03.012. Epub 2013 Apr 22. French. PMID 23618743